CLINICAL TRIAL: NCT06187922
Title: Effect of Perioperative Oral Pregabalin in Total Knee Replacement for Postoperative Pain
Brief Title: Effect of Perioperative Oral Pregabalin in Total Knee Replacement
Acronym: TKR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bahrain Defence Force Hospital (Other)
Responsible Party: Principal Investigator, Mehtash butt, Chief resident, Bahrain Defence Force Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BDF/R&REC/2023/674; BDF/R&REC/2023/674 (Other: crown prince training and research centre, Bahrain)
Record Dates: First submitted 2023-12-05; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Postoperative Pain
Keywords: Total knee replacement; Postoperative pain; Pregabalin; Adductor canal block; Dexmedetomidine
MeSH Terms: conditions — Pain, Postoperative | interventions — Pregabalin; Capsules

STUDY DESIGN:
Intervention Model Description: The patients will be randomly assigned into two equal groups; Group P: Pregablain group and Group C: control group. Group P will receive oral capsule pregabalin 75mg one hour preoperatively and will continue as B.D for 72 hrs, Group C will not receive any premedication preoperatively.
  Intraoperatively both groups will receive inj. Midazolam 2 mg before subarachnoid block with hyperbaric Bupivacaine 0.5% 2.5-3ml and fentanyl 15mcg in the operation theatre (OT). Both groups will also receive parecoxib 40mg IV and paracetamol 1G Intravenous (IV) as part of multimodal analgesia. Both groups will receive dexamethasone 8mg IV prophylactically. Postoperatively both groups will receive adductor canal block with bupivacaine and dexmedetomidine.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregabalin group (Active Comparator): this group of patient will receive cap pregabalin 75mg as premedication and will continue as twice daily dose for 72 hrs.
  Interventions: Drug: Pregabalin 75mg; Procedure: adductor canal block
- Control group (Sham Comparator): This group of patient will not receive cap pregabalin but it will receive standard medical care as routine
  Interventions: Procedure: adductor canal block

INTERVENTIONS:
Drug: Pregabalin 75mg — Group pregabalin will receive cap pregabalin 75mg as premedication and will continue as B.D dose for 72 Hrs.
  Other Names: capsule
  Arms: Pregabalin group
Procedure: adductor canal block — Both group will receive ultrasound guided Adductor canal block with bupivacaine 0.2% 20-30ml and dexmedetomidine 1mcg/Kg
  Other Names: peripheral nerve block

SUMMARY:
This interventional randomized control trial aim to determine efficacy and safety of Oral pregabalin in improving after surgery pain control in patients undergoing total knee replacement surgeries under regional anesthesia. We'll compare the efficacy of pregabalin between two groups, pregabalin group and control group on the basis of their opioid consumption after knee operation.

DETAILED DESCRIPTION:
After obtaining approval from the institutional ethical committee and informed written consent, 120 patients fulfilling the inclusion criteria will be included in this study. The patients will be randomly assigned into two equal groups; Group P: Pregabalin group and Group C: control group. Group P will receive oral capsule pregabalin 75mg one hour preoperatively and Group C will not receive any premedication preoperatively.

Intraoperatively both groups will receive inj. Midazolam 2 mg before subarachnoid block with hyperbaric Bupivacaine 0.5% 2.5-3ml and fentanyl 15mcg in the operation theatre (OT). Both groups will also receive parecoxib 40mg IV and paracetamol 1G Intravenous (IV) as part of multimodal analgesia. Both groups will receive dexamethasone 8mg IV prophylactically.

Postoperatively both groups will receive Ultrasound guided Adductor canal saphenous Nerve block in the PACU with 0.2% Bupivacaine 20-30ml & dexmeditomidine1.0mcg/kg. Group P will receive oral capsule pregabalin 75 mg Q12hourly from the 1st dose for next 60 hours. Group C will not receive any medication. Both groups will receive paracetamol 1G IV Q6Hourly and Rescue Analgesia will be provided with oral oxycodone 5mg TDS and Morphine PCA, in escalating manner as per patient requirement.

for 24 hrs. After 24 hours Both groups with receive tab paracetamol1 g Q4hourly, ibuprofen 400 Q8hourly along with Tab oxycodone as PRN Q8Hourly and PCA morphine.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 85 year
2. Elective Regional anesthesia.
3. Able to follow study protocol

Exclusion Criteria:

1. ASA -IV
2. Age <18 & > 85 years
3. Patients on pregabalin for chronic neuropathic pain.
4. Patient under General anesthesia
5. Patients with chronic liver failure
6. Patients with chronic renal failure on Hemodialysis
7. Patients on opioid (>3 month)
8. Patient with complicated knee surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale Score (0-10) | 72 hours
  visual analogue scale score at 4 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, 60 hours and 72 hours. minimum score mean good outcome

SECONDARY OUTCOMES:
Richmond Agitation Sedation Scale score {(+4) -0- (-5)} | 72 hours
  Richmond Agitation Sedation Scale score at 4 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, 60 hours and 72 hours. score +/-1 to 0 means good outcome.
Visual Analogue Sedation score at 1st Continuous Passive Movement | with in 24 hours
  visual analogue score at 1st continuous passive movement
Time of 1st analgesia request | within 24 hours
  Estimation of time for 1st complaint of pain
Incident of bradycardia | within 24hours
  Incident of reduction in Heart rate in 1st 24 Hours
Incident of Hypotension | within 24 hours
  Incident of reduced blood pressure below baseline
Total opioid consumption | within 72 hours
  Total opioid consumption in 72hours: Oxycodone/Morphine
Patient satisfaction | within 72 hours
  Patient satisfaction at 72 hours: rated as numeric 1-5 (1=not satisfied, 5=fully satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Al Muharraqi, FRCS,FDSRCS, Study Chair — Bahrain Defence Forces Hospital
Locations (1):
- Bahrain Defence Force, Manama, Bahrain

IPD SHARING:
Plan to Share IPD: No
We're still formulating the extended contact plan to follow patients for chronic pain.

REFERENCES:
- [Result] Li JW, Ma YS, Xiao LK. Postoperative Pain Management in Total Knee Arthroplasty. Orthop Surg. 2019 Oct;11(5):755-761. doi: 10.1111/os.12535. PMID 31663286
- [Result] Hah JM, Bateman BT, Ratliff J, Curtin C, Sun E. Chronic Opioid Use After Surgery: Implications for Perioperative Management in the Face of the Opioid Epidemic. Anesth Analg. 2017 Nov;125(5):1733-1740. doi: 10.1213/ANE.0000000000002458. PMID 29049117
- [Result] Attal N, Cruccu G, Baron R, Haanpaa M, Hansson P, Jensen TS, Nurmikko T. EFNS guidelines on the pharmacological treatment of neuropathic pain: 2010 revision. Eur J Neurol. 2010 Sep;17(9):1113-e88. doi: 10.1111/j.1468-1331.2010.02999.x. Epub 2010 Apr 9. PMID 20402746
- [Result] Ziyaeifard M, Mehrabanian MJ, Faritus SZ, Khazaei Koohpar M, Ferasatkish R, Hosseinnejad H, Mehrabanian M. Premedication with oral pregabalin for the prevention of acute postsurgical pain in coronary artery bypass surgery. Anesth Pain Med. 2015 Jan 17;5(1):e24837. doi: 10.5812/aapm.24837. eCollection 2015 Feb. PMID 25830118
- [Result] Chen YK, Boden KA, Schreiber KL. The role of regional anaesthesia and multimodal analgesia in the prevention of chronic postoperative pain: a narrative review. Anaesthesia. 2021 Jan;76 Suppl 1(Suppl 1):8-17. doi: 10.1111/anae.15256. PMID 33426669
- [Result] Sun Q, Liu S, Wu H, Ma H, Liu W, Fang M, Liu K, Pan Z. Dexmedetomidine as an Adjuvant to Local Anesthetics in Transversus Abdominis Plane Block: A Systematic Review and Meta-analysis. Clin J Pain. 2019 Apr;35(4):375-384. doi: 10.1097/AJP.0000000000000671. PMID 30475260
- [Result] Andersen JH, Jaeger P, Grevstad U, Estrup S, Geisler A, Vilhelmsen F, Dahl JB, Laier GH, Ilfeld BM, Mathiesen O. Systemic dexmedetomidine is not as efficient as perineural dexmedetomidine in prolonging an ulnar nerve block. Reg Anesth Pain Med. 2019 Mar;44(3):333-340. doi: 10.1136/rapm-2018-100089. Epub 2019 Jan 23. PMID 30679332
- See also: Pregabalin — http://reference.medscape.com/drug/lyrica-cr-pregabalin-343368

DOCUMENTS (2):
  • Study Protocol (2023-08-08): https://cdn.clinicaltrials.gov/large-docs/22/NCT06187922/Prot_000.pdf
  • Informed Consent Form (2023-02-19): https://cdn.clinicaltrials.gov/large-docs/22/NCT06187922/ICF_001.pdf